CLINICAL TRIAL: NCT02924311
Title: A Prospective Observational Study Conducted in France to Describe Routine Clinical Practice for Treatment naïve or Previously Treated Patients With Diabetic Macular Edema (DME) Who Are Starting IVT Aflibercept
Brief Title: Routine Clinical Practice for Use of Intravitreal Aflibercept Treatment in Patients With Diabetic Macular Edema
Acronym: APOLLON
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 18636
Record Dates: First submitted 2016-09-05; First posted 2016-10-05 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Previously treated patient: Already treated with any other treatment such as an anti-VEGF agent (other than IVT aflibercept), macular laser photocoagulation (laser), intravitreal steroid injection or implant (steroids) and initiating treatment with IVT aflibercept
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- Naïve patient: Not previously treated with an anti-VEGF agent, macular laser photocoagulation (laser) or intravitreal steroid injection or implant (steroids) and initiating treatment with IVT aflibercept
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- Entire study population: Already treated patient with any other treatment such as an anti-VEGF agent (other than intravitreal aflibercept), macular laser photocoagulation, intravitreal steroid injection and initiating treatment with intravitreal aflibercept and not previously treated patients with an anti-VEGF agent, macular laser photocoagulation or intravitreal steroids injection and initiating treatment with intravitreal aflibercept
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Eylea 40 mg/mL - recommended dose of 2 mg - intravitreal injection monthly for five consecutive months, which constitutes the loading dose. The loading dose is followed by one injection every two months. After 12 months of treatment, the interval between two injections can be prolonged or adapted according to visual and anatomical results.

SUMMARY:
The main objectives of this observational study were to describe outcomes, monitoring and treatment patterns of patients with diabetic macular edema in routine clinical practice who are either treatment naïve patients or previously treated patients. The total study population was evaluated as well as the two subgroups (previously treated patients and treatment naïve patients).

This study was designated to answer French Health Authority (HAS Haute Autorité de Santé) requirements.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 years or older
* Patient diagnosed with a visual impairment due to diabetic macular disease (as defined by HAS (Haute Autorité de Santé) recommendation).
* Patients in whom a decision to treat with intravitreal aflibercept has been made independently of the patient enrollment in the study
* Patient diagnosed with type 1 or 2 diabetes mellitus
* Patient who has been given appropriate information about the study and who has given his/her written, informed consent

Exclusion Criteria:

* Patient with other retinal disease at the time of inclusion
* Patients currently being treated with intravitreal aflibercept. This study will only include patients new to intravitreal aflibercept
* Systemic use of any anti / pro VEGF therapy (VEGF: Vascular Endothelial Growth Factor)
* Patient taking part in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment naïve and previously treated diabetic macular disease patients initiating a treatment with intravitreal aflibercept.
  The prescription of the medicines is clearly separated from the decision to include the patient in the study
Sampling Method: Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Mean change in Best Corrected Visual Acuity from baseline to month 12 in treatment naïve patients and previously treated patients | At baseline and 12 months

SECONDARY OUTCOMES:
Mean change in Best Corrected Visual Acuity between baseline and 12-month follow-up for the entire study population | At baseline and 12 months
Mean change in Best Corrected Visual Acuity between baseline and 24-month follow-up for all groups | At baseline and 24 months
Mean change in Central Retinal Thickness between baseline and 12-month follow-up for all groups | At baseline and 12 months
Mean change in Central Retinal Thickness between baseline visit and 24-month follow-up for all groups | At baseline and 24 months
Type of the previous treatment(s) in previously treated patients | At baseline
  i.e: photocoagulation laser therapy, anti-VEGF treatment, intraocular steroids
Duration (months) of the previous treatment in previously treated patients | At baseline
Date of the last administered treatment in previously treated patients | At baseline
Reason for starting intravitreal aflibercept | At baseline, 12 months and 24 months
  i.e: clinically significant macular edema conducting to a decrease of visual acuity, early care of DME, laser photocoagulation or vitrectomy not indicated, diabetes care not optimized
Number of eyes injected | Up to 24 months
Number of visits with injection | Up to 24 months
Interval (days) between injections | Up to 24 months
Type of adjunctive therapy post IVT aflibercept initiation | Up to 24 months
  i.e: surgery, focal laser, steroids, etc
Proportion of patients with change in fluorescein angiograph outcomes between baseline and 24-month follow-up for all groups | At baseline and 24 months
Proportion of patients with change in fundus photography outcomes between baseline and 24-month follow-up for all groups | At baseline and 24 months
Proportion of patients with no fluid determined by optical coherence tomography (OCT) between baseline and 24-month follow-up | At baseline, 12 months and 24 months
Mean change in HbA1c level during macular disease monitoring | At baseline, 12 months and 24 months
  HbA1c: Glycated haemoglobin A1c
Mean change in blood pressure during macular disease monitoring | At baseline, 12 months and 24 months
Duration of the disease (DME Monitoring) | At baseline
Number of visits for monitoring only (DME Monitoring) | Up to 24 months
Number of visits for injection only (DME Monitoring) | Up to 24 months
Number of visits combining monitoring and injection (DME Monitoring) | Up to 24 months
Number of monitoring visits for diabetes (by diabetologists, general practitioners) outside the study center over 12 and 24 months (if known by the ophthalmologist) (DME monitoring) | Up to 24 months
  Monitoring visits for diabetes by diabetologists or general practitioners outside the study center
Number of visits with OCT assessments (DME monitoring) | Up to 24 months
Number of visits with fundus photography assessments (DME monitoring) | Up to 24 months
Number of visits with fluorescein angiography assessments (DME monitoring) | Up to 24 months
Number of visits with visual acuity measurements (DME monitoring) | Up to 24 months
Number of participants with ocular and non-ocular safety events | Up to 24 months

OTHER OUTCOMES:
Number of prior treatments (DME Monitoring) | Up to 24 months
Number of patients with prior photocoagulation laser therapy (DME Monitoring) | Up to 24 months
Number of patients with prior anti-VEGF treatment (DME Monitoring) | Up to 24 months
Number of patients with prior intraocular steroids (DME Monitoring) | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, France

REFERENCES:
- [Result] Korobelnik JF, Daien V, Faure C, Tadayoni R, Giocanti-Auregan A, Dot C, Kodjikian L, Massin P; APOLLON study investigators. Two-year outcomes of the APOLLON observational study of intravitreal aflibercept monotherapy in France in patients with diabetic macular edema. Sci Rep. 2022 Oct 29;12(1):18242. doi: 10.1038/s41598-022-22838-1. PMID 36309572
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/